CLINICAL TRIAL: NCT01729312
Title: Pilot Study to See if There is a Improvement in Landing Techniques After a 9 Week Strenghtening Program, Which May Decrease ACL Tears in Female Athletes
Brief Title: Female Acl Prevention Study Where we Look at Landing Techniques Pre/Post Nine Week Strenghtening Program
Status: Terminated | Type: Observational
Why Stopped: Not enough participants to validate study.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Maria Blokdijk, certified athletic trainer, Henry Ford Health System
Other Study IDs: female acl prevention study
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Prevention of ACL Thru Strengthening Program

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens are taken
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To make reading this consent form easier, the word "participant" refers to you or your child (if a minor) throughout the consent form. This research is being done to study the effects of an eighteen-session strengthening program and to see if there is a relationship between the female athletes improving their landing techniques which has been proven to decrease anterior cruciate ligament injuries.

Participants have been asked to take part in a research study because you are a female athlete involved in a sport that has an increased anterior cruciate ligament injury rate. The purpose of this research study is to find out if an eighteen-session strengthening program will decrease your anterior cruciate ligament injury rate.

There will be approximately ninety-four (94) people in this research study at Henry Ford Health System (HFHS).

DETAILED DESCRIPTION:
The purpose of this research program is to use Dartfish technology and Functional Movement Screen to assess female athletes pre- and post injury prevention program.The study will include ninety-four females: forty-seven who complete a nine week program focusing on neuromuscular and proprioceptive exercises to improve landing techniques, and forty-seven who go about their normal preseason training regimen. This program has no more risk than if each athlete were to work out at their own gym. Each athlete will be given two questionnaires before and after completing the program in order to determine their level of activity has changed as well as uncover any underlying knee issues. Participants will also go through a series of functional and movement tests to reveal any imbalances, and determine whether or not they have improved by going through the prevention program.

All functional and movement tests will be video recorded. These recordings will only be used for the purpose of conducting this research study and will only be viewed by the HFHS investigators participating in the study. We will follow-up with each athlete one year later to see if there are any lasting effects from the program and re-test each athlete at that time to validate any results

ELIGIBILITY:
Inclusion Criteria:females only age 13-16 -

Exclusion Criteria:all males females younger than 13 and older than 16

-

Ages: 13 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: female athletes in age of 13-16
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy High School, Farmington, Michigan, United States

IPD SHARING:
Plan to Share IPD: No